CLINICAL TRIAL: NCT05149989
Title: Proning Pillows for Intensive Care Unit: Comparison of Chest and Pelvis Interface Pressure Distributions Between a Novel Proning Pillow System and Standard Pillows in Healthy Subjects
Brief Title: Comparison Between a Novel Proning Pillow System and Standard Pillows
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SP0857
Record Dates: First submitted 2021-11-23; First posted 2021-12-08 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2022-06

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proning (Experimental): Proned on standard and proning pillows
  Interventions: Device: Proning Pillow System

INTERVENTIONS:
Device: Proning Pillow System — Participants will be asked to lie on the proning pillows in prone position for no more than 5 minutes. Each participant will then be asked to lie on standard hospital pillows for no more than 5 minutes.

SUMMARY:
During the COVID-19 pandemic, intensive care units (ICUs) across the country have been inundated with increasing numbers of COVID patients. Hypoxic patients in ICU require mechanical ventilation and this can be improved by proning these patients to improve oxygenation and prevent ventilator-induced lung injury. Standard practice is to use standard hospital pillows to support the pelvis and chest of the patient while they are proned. These pillows do not provide much support to the patients and often need to be adjusted due to the patient 'sinking' into them. Prolonged pronation also leads to pressure sores in these anatomical locations which burden the Trust financially and also cause distress to patients.

A new proning pillow system was developed by Dr Sashika Selladurai and manufactured for the ICU in Aintree hospital which is made from polyurethane memory foam designed to relieve pressure on the patients and prevent pressure sores that often occur during prolonged proning. The pillow system is also designed to withstand the load of heavier patients and reduce the risk of 'sinking' into the pillows when proned for long periods of time.

The aim of the study is to compare the performance of the new proning pillow system with standard pillows, particularly in relation to the risk of pressure sores, by evaluating differences in chest and pelvis interface pressures between the two pillow types. This will be done by having healthy NHS staff lie on the pillows in the prone position for a short period of time while recording the pressure distribution on the pillows using pressure mats placed between them and the pillows. This will help understand the relative risk of pressure sores developing when the new pillow system is used. It is hypothesised that the new pillow system does not increase the risk of pressure sores developing.

The new proning pillow system is a Class 1 CE marked medical device. The proning pillow system consists of a chest pillow and a pelvis pillow made from memory foam designed to reduce contact pressures and peak interface pressures in patients and allow patients to be placed in neutral position for ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Work for Liverpool University Hospital NHS Foundation Trust
* Participant is willing and able to give informed consent for participation in the study.
* Agree to have weight, height, chest and waist measurements taken
* Agree to the study protocol
* Aged 18 years or above.

Exclusion Criteria:

* Presentation of skin lesions
* Absence of any limb
* Female participant who is pregnant
* Have a lower back problem
* Pain or injury in shoulders or arms
* History of conditions that would make it difficult to lie prone, such as pressure injury or surgery within six months leading up to the study
* Any conditions that significantly affect movement and sensation such as diabetes or mobility limitations

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proning
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: NHS staff
Arm/Group | Proning
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 50

OUTCOME MEASURES:

1. Primary Outcome: Peak Chest and Pelvis Interface Pressures
Description: The maximum values of pressure measured by the two pressure mats, one placed in the chest region and on in the pelvis region, measured in mmHg.
Time Frame: 10 minutes
Population: Population was analysed in two separate groups: male (20) and female (30)
Measure: Mean (Inter-Quartile Range); unit: mmHg
Arm/Group | Proning
Number analyzed (Participants) | 50
mmHg
  Peak pressure: proning pillow, chest, male: number analyzed (Participants) | 20
  Peak pressure: proning pillow, chest, male | 88.1 [77.3 to 99.3]
  Peak pressure: standard pillow, chest, male: number analyzed (Participants) | 20
  Peak pressure: standard pillow, chest, male | 71.5 [59.0 to 72.2]
  Peak pressure: proning pillow, chest, female: number analyzed (Participants) | 30
  Peak pressure: proning pillow, chest, female | 69.6 [61.9 to 78.8]
  Peak pressure: standard pillow, chest, female: number analyzed (Participants) | 30
  Peak pressure: standard pillow, chest, female | 64.3 [59.7 to 74.4]
  Peak pressure: proning pillow, pelvis, healthy males: number analyzed (Participants) | 6
  Peak pressure: proning pillow, pelvis, healthy males | 70.4 [53.6 to 84.7]
  Peak pressure: standard pillow, pelvis, healthy males: number analyzed (Participants) | 6
  Peak pressure: standard pillow, pelvis, healthy males | 40.2 [35.3 to 44.9]
  Peak pressure: proning pillow, pelvis, overweight males: number analyzed (Participants) | 14
  Peak pressure: proning pillow, pelvis, overweight males | 96.3 [82.0 to 107.2]
  Peak pressure: standard pillow, pelvis, overweight males: number analyzed (Participants) | 14
  Peak pressure: standard pillow, pelvis, overweight males | 47.1 [39.8 to 54.0]
  Peak pressure: proning pillow, pelvis, healthy females: number analyzed (Participants) | 19
  Peak pressure: proning pillow, pelvis, healthy females | 86.0 [68.2 to 94.4]
  Peak pressure: standard pillow, pelvis, healthy females: number analyzed (Participants) | 19
  Peak pressure: standard pillow, pelvis, healthy females | 45.5 [36.6 to 53.1]
  Peak pressure: proning pillow, pelvis, overweight females: number analyzed (Participants) | 11
  Peak pressure: proning pillow, pelvis, overweight females | 84.4 [68.7 to 94.4]
  Peak pressure: standard pillow, pelvis, overweight females: number analyzed (Participants) | 11
  Peak pressure: standard pillow, pelvis, overweight females | 45.0 [40.8 to 50.8]

ADVERSE EVENTS:
Time Frame: 10 minutes
Arm/Group | Proning
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT05149989/Prot_SAP_000.pdf